CLINICAL TRIAL: NCT01895244
Title: Highdose Chemotherapy and Transplantation of 34+ Selected Stem Cell for Progressive Systemic Sclerosis - Modification According to Manifestation
Brief Title: Autologous Stem Cell Transplantation for Progressive Systemic Sclerosis
Acronym: AST-MOMA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Joerg Henes, Dr. med. Joerg Henes, University Hospital Tuebingen
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AST MOMA
Record Dates: First submitted 2013-07-01; First posted 2013-07-10 (Estimated); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Scleroderma; Cardiac Involvement; Autologous Stem Cell Transplantation
Keywords: scleroderma; autologous stem cell transplantation; thiotepa; cluster of differentiation (CD) 34 selection
MeSH Terms: conditions — Scleroderma, Diffuse | interventions — Antigens, Differentiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conditioning with CYC/ antithymocyte globulin (ATG) (Experimental): Each patient receives stem cell transplantation open label with cluster of differentiation (CD)34 selected stem cells mobilisation and conditioning depending on manifestation If cardiac manifestation: Conditioning with CYC 2 x 50mg + thiotepa 2x5mg + ATG If no cardiac manifestation: Conditioning with 4 x 50mg CYC + ATG
  Interventions: Drug: Autologous stemcell transplantation with CD (cluster of differentiation) 34 selected stem cells
- Conditioning with CYC/Thiotepa/ATG (Experimental): In patients with cardiac manifestations as defined in the protocol the conditioning for stem cell transplantation is changed to Cyclophosphamide (CYC), thiotepa and ATG
  Interventions: Drug: Autologous stemcell transplantation with CD (cluster of differentiation) 34 selected stem cells

INTERVENTIONS:
Drug: Autologous stemcell transplantation with CD (cluster of differentiation) 34 selected stem cells — If no active alveolitis: mobilisation with 2x1g Cyclophosphamide If active alveolitis: mobilisation with 2x1.5g Cyclophosphamid If cardiac manifestation: Conditioning with CYC 2 x 50mg + thiotepa 2x5mg + ATG If no cardiac manifestation: Conditioning with 4 x 50mg CYC + ATG

SUMMARY:
Autologous stem cell therapy has been shown to be effective in patients with systemic sclerosis. Nevertheless treatment is associated with treatment related mortality and patients die during follow up despite successful transplantation.

Intention of this trial is to improve overall survival by modifying the existing protocol used for the ASTIS trial.

To reduce treatment toxicity we reduce the dose of Cyclophosphamide (CYC) for mobilisation to 2x1g.

Especially in patients with cardiac manifestations we also modify the conditioning regimen by adding thiotepa and reducing CYC; as CYC has known cardiotoxic side effects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of progressive systemic sclerosis <7 years
* Progressive course despite cyclophosphamide pretreatment
* Cyclophosphamide i.v.: at least 3 x with 500-1000 mg/m² every 3-4 weeks or
* Cyclophosphamide p.o. with at least 100mg/day for at least 2 months or
* Contraindication to treatment with cyclophosphamide
* Progress defined as at least one of the following criteria:

  * Increase in the mRSS
  * Worsening of the lung function
  * Increase in fibrosis/alveolitis in thorax CT
  * Worsening kidney function through manifestation of systemic sclerosis
* Limited or diffuse cutaneous progressive form of Ssc with organ manifestation in the lungs/heart or kidneys

Exclusion Criteria:

* Age <18 years
* Pregnancy or inadequate contraception
* Severe heart failure with ejection fraction (EF) < 30% in echo
* Pulmonary arterial hypertension with systolic pulmonary arterial pressure (PAPsys) >50mm Hg
* Kidney insufficiency: creatinine clearance <30 ml/min
* Reduced lung function
* Inspiratory vital capacity (IVC) < 50% of normal
* Carbon monoxide (CO)-Diffusion capacity SB < 40%
* Previously damaged bone marrow
* Leukopenia < 2,000/µl
* Thrombopenia < 100,000/µl
* Previous myelotoxic treatment:
* Cyclophosphamide > 50g cumulative (relative)
* Infection (Hepatitis B/C, HIV, Salmonella carrier, syphilis, relative: history of tuberculosis)
* Severe concomitant psychiatric illness (depression, psychosis)
* Substance dependence
* Continued nicotine abuse
* Continued alcohol abuse
* Continued drug abuse
* Consent not given
* Poor compliance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2021-09 (Actual); Study Completion 2024-06 (Actual)

PRIMARY OUTCOMES:
Efficay - Overall survival | 3 years
  Number of patients that are alive after 3 years

SECONDARY OUTCOMES:
Safety - Treatment related mortality | 100 days
  Treatment related mortality: number of patients who die during the first 100 days after transplantation
Time to engraftment | 2 months
  Time in days from day 0 to platelet count > 20.000 and granulocytes >500/µl
Progression free survival | 3 years
  Time after transplantation without symptoms of disease activity
Efficacy - Lung function test and Skin | 3 years
  Number of patients that achieve either improvement of >25% in mRSS or > 10% in FVC or DLCO

OTHER OUTCOMES:
Efficacy - Patient reported outcome | 3 years
  Differences in Health Assessment Questionnaire (HAQ)

CONTACTS AND LOCATIONS:
Overall Officials: Joerg C Henes, MD, Principal Investigator — University Hospital Tuebingen, Department of oncology, hematology, rheumatology
Locations (1):
- University Hospital Tuebingen; Department of oncology, hematology, rheumatology, immunology and pulmology, Tübingen, Germany

REFERENCES:
- [Derived] Henes JC, Koetter I, Horger M, Schmalzing M, Mueller K, Eick C, Bauer A, Vogel W, Kanz L. Autologous stem cell transplantation with thiotepa-based conditioning in patients with systemic sclerosis and cardiac manifestations. Rheumatology (Oxford). 2014 May;53(5):919-22. doi: 10.1093/rheumatology/ket464. Epub 2014 Jan 22. PMID 24459219